CLINICAL TRIAL: NCT00498147
Title: Does Managed Diabetes Care Decrease Cardiovascular Complications of Diabetes?
Brief Title: Determining Rates of Cardiovascular Complications Among Patients of a Managed Diabetes Care Program
Acronym: DECIDE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Group Health Centre (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Silvana Spadafora, Group Health Centre
Other Study IDs: DECIDE
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Disease Management; Diabetes Complications; Diabetic Vascular Complications; Diabetic Neuropathy; Diabetic Nephropathy; Diabetic Retinopathy
Keywords: amputation; angina; angiography; angioplasty; arterial disease; artery disease; bypass; CABG; cad; carotid; cerebral accident; CHF; CRF; CVA; endarterectomy; heart attack; heart failure; infarct; kidney disease; kidney failure; laser; nephropathy; neuropathy; pad; PCI; percutaneous coronary; percutaneous transluminal; pvd; renal failure; retinopathy; revascularization; schemia; stenosis; stent; stroke; transient; ulcer; vascular disease
MeSH Terms: conditions — Diabetes Complications; Diabetic Angiopathies; Diabetic Neuropathies; Diabetic Nephropathies; Diabetic Retinopathy; Angina Pectoris; Coronary Artery Disease; Stroke; Myocardial Infarction; Heart Failure; Infarction; Kidney Diseases; Renal Insufficiency; Peripheral Vascular Diseases; Retinal Diseases; Constriction, Pathologic; Ulcer; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADEC <6months: Patients new to the ADEC program who will be provided the ADEC interventions (prospective study)
  Interventions: Other: ADEC Program
- ADEC >6months: Patients who have been with the ADEC program as early as 2002 (coincides with ADEC's EMR initiation date) who continue to be provided the ADEC interventions (combined retrospective/prospective study)
  Interventions: Other: ADEC Program

INTERVENTIONS:
Other: ADEC Program — Interventions (managed diabetes care) employed by the ADEC Program include: diabetes education, nutrition care, individual and group counseling sessions, foot care, and insulin and oral diabetes medication adjustments with a signed medical directive. ADEC Diabetes Educators (Registered Dietitians and Registered Nurses) will use adult education principles throughout the education process and promote self-care by encouraging responsibility and promoting a positive attitude towards acceptance of diabetes. All patients will be encouraged to self-monitor their blood glucose at home. Team member collaboration and with other agencies to promote a total client care approach to diabetes management will be employed.
  Other Names: Managed Diabetes Care

SUMMARY:
The primary objective of this study is to identify whether cardiovascular complication rates are lower in patients who participate in managed diabetes care, in comparison to provincial and national rates. This study will involve an electronic medical record (EMR) chart audit, augmented by a manual review of hospital and other pertinent medical records, as necessary.

DETAILED DESCRIPTION:
The DECIDE study will identify whether cardiovascular complication rates (the composite rate of myocardial infarction (MI), Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Grafting (CABG), stroke, carotid endarterectomy, peripheral revascularization, and peripheral amputation) are lower in patients who participate in managed diabetes care by ADEC in comparison to provincial and national rates. Comparison statistics will be provided by the Institute of Evaluative Sciences (ICES) Atlas 2003 and other Diabetes studies such as the 2005 DICE study. Complications such as nephropathy and retinopathy will be documented, along with hospitalization rates and all cause mortality. Clinical outcomes relevant to diabetes management such as blood pressure and lipids will also be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory patients over the age of 18 years with diabetes mellitus.
2. Current enrolment in ADEC program (>6 months)or new enrolment in ADEC program (<6 months).
3. Confirmed diagnosis of diabetes mellitus, according to the current Canadian Diabetes Guidelines.
4. Informed consent provided

Exclusion Criteria:

1. History of only gestational diabetes.
2. Non-GHC member.
3. GHC patients with diabetes who do not attend the ADEC program.
4. Unable to give informed consent.
5. Any conditions/circumstances that prevent the patient from attending ADEC sessions or participating fully in the program.
6. Refusal to allow research staff access to medical records, including hospital charts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients of the Group Health Centre who are over the age of 18 years with a confirmed diagnosis of diabetes mellitus and who are enrolled in the Algoma Diabetes Education and Care (ADEC) program. ADEC is a managed diabetes care program and part of the Group Health Centre (GHC), a multi-specialty, interdisciplinary, ambulatory care facility located in Sault Ste. Marie, a northern Ontario community. With diagnostic services and a comprehensive electronic medical record, GHC provides health care to most of the community's population of approximately 75,000.
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Rates of cardiovascular events and other complications of diabetes compared to provincial and national rates | 1 year

SECONDARY OUTCOMES:
The secondary outcomes will be total mortality, CV- related events, and other selected complications of diabetes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Spadafora, MD FRCPC, Principal Investigator — The Group Health Centre
Locations (1):
- Group Health Centre, Sault Ste. Marie, Ontario, Canada

REFERENCES:
- See also: Group Health Centre website — http://www.ghc.on.ca